CLINICAL TRIAL: NCT02555982
Title: Evaluation of Botulinum Toxin Injection Efficacy in the Treatment of Head Essential Tremor by a Multi-center, Randomized, Double-Blind, Parallel-group, Placebo-controlled Study
Brief Title: Evaluation of Botulinum Toxin Injection Efficacy in the Treatment of Head Essential Tremor
Acronym: Btx-HT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0245; 2015-000162-59 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-22 (Estimated); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Essential Head Tremor
Keywords: Essential Head tremor; Botulinum toxin injections; Quality of life; Embarrassment assessment

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Patients eligible for inclusion will be randomized to one of the two groups:
  * Experimental group: 60 patients will receive 2 injections of Btx A (BOTOX - Allergan), one on D0 and one at 12W (into each splenius capitis).
  * Control group: 60 patients will receive 2 injections of placebo, one on D0 and one at 12W (into each splenius capitis).
  Interventions: Drug: BOTOX ® 200 Unités
- CONTROL GROUP (Other): Patients eligible for inclusion will be randomized to one of the two groups:
  * Experimental group: 60 patients will receive 2 injections of Btx A (BOTOX - Allergan), one on D0 and one at 12W (into each splenius capitis).
  * Control group: 60 patients will receive 2 injections of placebo, one on D0 and one at 12W (into each splenius capitis).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOTOX ® 200 Unités — Patients eligible for inclusion will be randomized to one of the two groups:
  * Experimental group: 60 patients will receive 2 injections of Btx A (BOTOX - Allergan), one on D0 and one at 12W (into each splenius capitis).
  * Control group: 60 patients will receive 2 injections of placebo, one on D0 and one at 12W (into each splenius capitis).
  Arms: EXPERIMENTAL GROUP
Drug: Placebo — Control group: 60 patients will receive 2 injections of placebo, one on D0 and one at 12W (into each splenius capitis).
  Arms: CONTROL GROUP

SUMMARY:
Essential head tremor (HT) does not usually respond to drug treatment such as propranolol or primidone or to surgical treatment such as deep brain stimulation of the thalamic ventralis intermedius nucleus. Botulinum toxin (Btx) is widely used and efficient in the treatment of blepharospasm and cervical dystonia. Btx prevents the release of acetylcholine in synapses, leading to a reduction of pathological muscle movement. Very little information is available on its efficacy on HT. Two published reports suggested that local Btx A injections could be an effective and safe approach for treating HT. Given the scarcity of published data (small samples, open studies, different doses of Btx used, heterogeneous populations, several muscles injected, etc.), the aim of this study is to demonstrate the efficacy of Btx injections in essential HT by a multi-center, randomized, double-blind, parallel-group, placebo-controlled study.

Principal objective: To evaluate the efficacy of botulinum toxin injections in the treatment of head tremor.

Secondary objectives:

* - To evaluate the tolerance of botulinum toxin injections in the treatment of head tremor.
* - To evaluate the impact of botulinum toxin injections on the patients' quality of life and embarrassment.
* To evaluate the changes of tremor characteristics induced by a Btx treatment using a 3D accelerometer wireless portable system (Xsens MTw wireless motion tracker system) (tremor frequency, tremor displacement, mean peak amplitude, distance traveled) and a new video system device to analyze head tremor characteristics

DETAILED DESCRIPTION:
Type of study: multi-center, randomized, double-blind, parallel-group, placebo-controlled therapeutic clinical trial.

Number of centers: 19 centers : Clermont-Ferrand, Paris (Fondation Rothschild, APHP, Hôpital Lariboisière, Hôpital Avicenne de Bobigny), Toulouse, Lyon, Amiens, Bordeaux, Narbonne, Lille, Strasbourg, Nîmes, Marseille, Besançon, Aix, Montpellier, Pau,Poitiers

Medical product Botulinum toxin type A, 200U (BOTOX ® 200 Unités, Allergan)

Patients

Patients eligible for inclusion will be randomized to one of the two groups:

* Experimental group: 60 patients will receive 2 injections of Btx A (BOTOX - Allergan), one on D0 and one at 12W (into each splenius capitis).
* Control group: 60 patients will receive 2 injections of placebo, one on D0 and one at 12W (into each splenius capitis).

Study Performance Patients will be injected twice, with an interval of 12 weeks (D0 and 12W). On D0, patients will receive 75U of Btx A (BOTOX ® - Allergan) in each splenius capitis; at 12W, patients will receive the same dose as on D0 (if the first injection is effective according to the CGI- improvement by at least two points), or a higher dose (100U) (if the first injection is ineffective according to the CGI- non improvement or improvement by less than two points).

Patients will be assessed at baseline D0, 6 weeks (6W), 12 weeks (12W), 18 weeks (18W) and 24 weeks (24W) after D0 as follows:

Visit 1 (baseline):

* Signature of an informed consent form.
* Demographic and clinical characteristics (sex, age, disease duration, treatments).
* Clinical evaluation:
* Neurological evaluation: Fahn-Tolosa-Marin Tremor Rating Scale (TRS), Tsui Scale.
* The Quality of life in Essential Tremor (QUEST), the Essential Tremor Embarrassment Assessment (ETEA).
* Accelerometer recording and videotape recording.

Visits at 6W, 12W, 18W and 24W

* Clinical evaluation:
* TRS.
* CGI.
* QUEST / ETEA.
* Accelerometer recording and videotape recording.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a head tremor without (isolated) or with associated
* tremor in any other body parts.
* The HT must be troublesome for the patients (TRS 2 for the head tremor
* severity item).
* Patients never treated with botulinum toxin or not treated with botulinum toxin for this indication for at least 4 months.
* Men or women aged from 18 to 80 years old.
* Social security coverage.
* Ability to provide informed consent.

Exclusion Criteria:

* Patients with tremor from cerebellar syndrome (multiple sclerosis, etc.).
* Patients with a predominant dystonic jerky or myoclonic head tremor using
* the Tsui scale (>1).
* Oral treatments for HT are allowed but must be stable during the study.
* Any contra-indication to Botulinum toxin.
* Women without efficient contraception.
* Patients under supervision or (legal) guardianship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
clinical state improvement of patients evaluated by the Clinical Global Impression of Change (CGI) | at 18 weeks
  clinical state improvement of patients evaluated by the Clinical Global Impression of Change (CGI) (improvement by at least two points) measured 6 weeks after the 2nd injection of Btx (at 18W).
% of responders defined with CGI | at 6 weeks
% of responders defined with CGI | at 18 weeks
The Fahn-Tolosa-Marin Tremor Rating Scale (TRS) (sub item head) | at day 0
The Fahn-Tolosa-Marin Tremor Rating Scale (TRS) (sub item head) | at 6 weeks
The Fahn-Tolosa-Marin Tremor Rating Scale (TRS) (sub item head) | at 12 weeks

SECONDARY OUTCOMES:
The Fahn-Tolosa-Marin Tremor Rating Scale (TRS) (sub item head) | at 18 weeks
The Fahn-Tolosa-Marin Tremor Rating Scale (TRS) (sub item head) | at 24 weeks
The Essential Tremor Embarrassment Assessment (ETEA) | at day 0
The Essential Tremor Embarrassment Assessment (ETEA) | at 6 weeks
The Essential Tremor Embarrassment Assessment (ETEA) | at 12 weeks
The Essential Tremor Embarrassment Assessment (ETEA) | at 18 weeks
The Essential Tremor Embarrassment Assessment (ETEA) | at 24 weeks
The Quality of life in Essential Tremor (QUEST) | at day 0
The Quality of life in Essential Tremor (QUEST) | at 6 weeks
The Quality of life in Essential Tremor (QUEST) | at 12 weeks
The Quality of life in Essential Tremor (QUEST) | at 18 weeks
The Quality of life in Essential Tremor (QUEST) | at 24 weeks
tremor frequency measured by accelerometer | at day 0
tremor frequency measured by accelerometer | at 6 weeks
tremor frequency measured by accelerometer | at 12 weeks
tremor frequency measured by accelerometer | at 18 weeks
tremor frequency measured by accelerometer | at 24 weeks
mean peak amplitude measured by accelerometer | at day 0
mean peak amplitude measured by accelerometer | at 6 weeks
mean peak amplitude measured by accelerometer | at 12 weeks
mean peak amplitude measured by accelerometer | at 18 weeks
mean peak amplitude measured by accelerometer | at 24 weeks
distance traveled measured by accelerometer | at day 0
distance traveled measured by accelerometer | at 6 weeks
distance traveled measured by accelerometer | at 12 weeks
distance traveled measured by accelerometer | at 18 weeks
distance traveled measured by accelerometer | at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franck Durif, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (17):
- France (17):
  - Centre Hospitalier Pays D'Aix, Aix-en-Provence
  - CHU d'Amiens, Amiens
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Haut-Levêque, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital R Salendro, Lille
  - Hôpital neurologique, Lyon
  - Hôpital de la Timone, Marseille
  - CH Narbonne, Narbonne
  - Hôpital Caremeau, Nîmes
  - AP-HP, Paris
  - Fondation Rothschild, Paris
  - Hopital Lariboisière, Paris
  - Hôptal Avicenne de Bobigny, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital de Hautepierre, Strasbourg
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Marques A, Pereira B, Simonetta-Moreau M, Castelnovo G, De Verdal M, Fluchere F, Laurencin C, Degos B, Tir M, Kreisler A, Blanchet-Fourcade G, Guehl D, Colin O, Poujois A, Sangla S, Tatu L, Derost P, Gayraud D, Tranchant C, Amarantini D, Devos D, Rascol O, Corvol JC, Durif F, Rieu I; Btx-HT Study Group. Trial of Botulinum Toxin for Isolated or Essential Head Tremor. N Engl J Med. 2023 Nov 9;389(19):1753-1765. doi: 10.1056/NEJMoa2304192. PMID 37937777